CLINICAL TRIAL: NCT04811157
Title: The Effect of Functional Dairy Products Enriched With Dietary Fibers on Human Health and Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Food and Fermentation Technologies (Other)
Collaborators: SYNLAB Eesti OÜ, Tallinn, Estonia (Unknown); AS FARMI Piimatööstus, Jõhvi, Estonia (Unknown)
Responsible Party: Principal Investigator, Madis Jaagura, Project Manager, Center of Food and Fermentation Technologies
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2014-2020.4.02.19-0198
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: microbiome; bifidobacteria; fermented dairy product
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Healthy adults consuming test product
  Interventions: Dietary Supplement: Test product
- Control group (Placebo Comparator): Healthy adults consuming control product
  Interventions: Dietary Supplement: Control product

INTERVENTIONS:
Dietary Supplement: Test product — 200 g/day of unsweetened yogurt supplemented with a dietary fiber blend
  Arms: Test group
Dietary Supplement: Control product — 200 g/day of unsweetened yogurt
  Arms: Control group

SUMMARY:
The purpose of this dietary intervention is to study the effects of dietary fibers on the gut microbiota and use yoghurt as the carrier.

Hypothesis 1: Intake of dietary fibers improves the blood lipid profile of the participants.

Hypothesis 2: Intake of dietary fibers stabilizes the gut microbiome (e.g., low diversity) of the participants, improves gut health and normalizes gastrointestinal function and bowel habits.

DETAILED DESCRIPTION:
The study design is a parallel randomized, prospective, pre-post intervention trial. The main goal of this study is to investigate the effect of the dietary fibers in an unsweetened yoghurt. Fermented dairy products have naturally a very low dietary fiber content, but such products can be supplemented with variety of dietary fibers and promote the growth of beneficial gut bacteria. Also, as fermented milk products contain live bacteria, it is possible that prebiotic fibers could support the growth of the starter-culture based strains in the human gut.

PRE-STUDY EVALUATION AND TESTING

1. Complete pre-study questionnaire
2. Complete orientation to the study and provide voluntary consent to join the study
3. Collection of coded intervention products, sampling supplies, and instructional materials 0-WEEK QUESTIONNAIRE AND LABORATORY VISIT

1. Record food intake and gastrointestinal function for 3 days 2. Collect health data and provide a 3-day food frequency questionnaire 3. Provide a stool and blood sample at the laboratory 2-WEEK QUESTIONNAIRE AND LABORATORY VISIT

1. Record food intake and gastrointestinal symptoms for 3 days
2. Collect health data and provide a 3-day food frequency questionnaire
3. Provide a stool and blood sample at the laboratory BLOOD SAMPLE ANALYSES

1. Provide the blood sample at the laboratory in the morning in an overnight fasted state.

DIETARY INTERVENTION

1. Daily intake of a test or control product for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-55
* Normal bowel function
* Regular consumer of dairy products, willing to consume dairy products daily for 2 weeks
* Ability to provide a signed written informed consent
* Willing to provide stool and blood specimens 2 times over the 2-week study period

Exclusion Criteria:

* Diagnosed history of chronic diseases including coronary heart disease, stroke, cancer, type 1 or 2 diabetes mellitus, inflammatory bowel disease, gastritis, autoimmune disease, or rheumatoid arthritis
* Medication: statins, blood pressure medications, antidepressants, other prescription medications
* History of bariatric operation, removal of the gallbladder.
* Food allergies, lactose intolerance
* Recent (previous 3 months) use of antibiotics
* Intake of highly dosed pre- or probiotics 2 weeks prior and during the study
* Current pregnancy or breastfeeding
* Volunteers showing previously unrecognized illness will also be excluded
* Individual unable to give informed consent

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the intestinal microbiota | 14 days
  Fecal microbiota analysis based on the 16S rRNA sequencing pre- and post-dietary intervention.
Evaluation of blood lipid profile | 14 days
  Triglycerides, total cholesterol, HDL-cholesterol, LDL-cholesterol pre- and post-dietary intervention in plasma (mmol/L).
Evaluation of blood glucose levels | 14 days
  Fasting glucose pre- and post-dietary intervention in plasma (mmol/L).

SECONDARY OUTCOMES:
Evaluation of the stool form | 14 days
  Stool form will be assessed using a validated 7-point scale called Bristol Stool Form Scale pre- and post-dietary intervention.
Evaluation of the defecation frequency | 14 days
  1. Evacuation frequency during 3 days pre- and post-dietary intervention.
  2. Evacuation frequency (number of bowel movements per week) pre- and post-dietary intervention.
Evaluation of the defecation timing | 14 days
  Evacuation timing 3 days before sampling pre- and post-dietary intervention.
Evaluation of the gastrointestinal symptoms | 14 days
  Frequency and severity of the gastrointestinal symptoms (Constipation, Diarrhea, Bloating, Flatulence, Cramps, Stomach pain). Scale of frequency: Never, Less than 10 times a year, Once a month, Once a week, Every day. Scale of severity: I do not have any gastrointestinal symptoms, Mild (does not disturb), Moderate, Strong (disturbs considerably).
Evaluation of the blood vitamin D status | 14 days
  25-OH vitamin D pre- and post-dietary intervention in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Madis Jaagura, MSc, Principal Investigator — TFTAK
Locations (1):
- Center of Food and Fermentation Technologies, Tallinn, Harju, Estonia

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized participant data could be made available for subsequent analysis in the mentioned institution (TFTAK).
  Data made public will include only aggregates or summaries of the collected data.

DOCUMENTS (1):
  • Informed Consent Form (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT04811157/ICF_000.pdf